CLINICAL TRIAL: NCT06641336
Title: Perceptions of Using RehAtt Mixed Reality System in Stroke Motor Rehabilitation
Brief Title: Perceptions of RehAtt Mixed Reality System
Acronym: RehAtt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: URIS202403
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: rehabilitation; mixed reality; motor rehabilitation; patients' perspective
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RehAtt (Experimental): Each patient was included in the introduction session (performed by a psychologist), three sessions of occupational therapy and three sessions of physiotherapy. Each session lasted for 30 minutes. Occupational-therapy training was focused on activities aimed at improving upper limb function; physiotherapy training was focused on balance, walking and standing.
  Interventions: Device: RehAtt

INTERVENTIONS:
Device: RehAtt — Each patient received the RehAtt intervention.

SUMMARY:
The study aims to explore the patients' perspective on usability and feasibility of the RehAtt™ mixed-reality system during upper limb, gait and balance function rehabilitation.

DETAILED DESCRIPTION:
Mixed reality is an immersive technology that can integrate virtual objects into the real world and adaptive scenarios. It offers the opportunity to train physical and cognitive aspects in stroke patients. The patients' perspectives were assessed with a semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* first ischaemic or hemorrhagic stroke,
* one-sided hemiparesis,
* adequate cognitive abilities.

Exclusion Criteria:

* severe cognitive impairment,
* aphasia,
* known presence of an epileptic seizure in the last year,
* other orthopaedic and neurological diseases affecting sensory or motor functions,
* inability to sit independently,
* severe visual impairment,
* severe depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interview | On the day of the end of the intervention
  The interview was based on a questionnaire that included rating-scale-based questions on mixed-reality therapy meeting the patient's needs, frustration during the exercise, ease of use, difficulties encountered, motivational aspect, likability and usefulness of each exercise, and open-ended questions on motivation, overall view of the mixed-reality system and possible unwanted effects.

CONTACTS AND LOCATIONS:
Overall Officials: Nataša Bizovičar, MD, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia